CLINICAL TRIAL: NCT01140334
Title: Maximizing Effectiveness of Integrated Treatment Approaches
Brief Title: Treatment for Psychological and Drug Abuse Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michael Kidorf, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1RC1DA028154-01 (NIH)
Record Dates: First submitted 2010-06-03; First posted 2010-06-09 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Substance Use Disorders
Keywords: Psychiatric adherence; Voucher incentives; Methadone treatment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reinforced On-Site Integrated Care (ROIC) (Experimental): Patients assigned to this condition will be treated at ATS for psychological problems. They will be scheduled to participate in individual therapy sessions with a psychiatrist and with their substance abuse counselor. They will also be referred to attend group therapy one time per week. In addition, they will be able to earn a voucher incentive for each week of psychiatric compliance.
  Interventions: Behavioral: Voucher Reinforcement
- Standard On-Site Integrated Care (SOIC). (Active Comparator): Patients assigned to this condition will be treated at ATS for psychological problems. They will be scheduled to participate in individual therapy sessions with a psychiatrist and with their substance abuse counselor. They will also be referred to attend group therapy one time per week.
  Interventions: Behavioral: Standard Control

INTERVENTIONS:
Behavioral: Voucher Reinforcement — Patients in this condition will be able to earn a voucher for each week that they have attended all scheduled psychiatric sessions. These sessions may include individual therapy appointments, group therapy appointments, or psychiatrist appointments. Each voucher will be worth $25, and can be exchanged for goods and services that will be purchased by a research assistant. The maximum amount of voucher earnings over the study is $300.
  Arms: Reinforced On-Site Integrated Care (ROIC)
Behavioral: Standard Control — Patients assigned to this condition will be treated at ATS for psychological problems. They will be scheduled to participate in individual therapy sessions with a psychiatrist and with their substance abuse counselor. They will also be referred to attend group therapy one time per week. No voucher incentive will be offered in this condition.
  Arms: Standard On-Site Integrated Care (SOIC).

SUMMARY:
The purpose of the study is to evaluate methods to help people in substance abuse treatment receive better psychiatric care. Patients enrolled in the study will be offered three months of standard psychiatric treatment, which consists of weekly individual counseling and group counseling, as well as regular appointments with a psychiatrist. Patients will be randomly assigned to standard psychiatric care or standard psychiatric care plus voucher incentives. These incentives can be earned by successfully attending all scheduled psychiatric appointments each week. The investigators expect that patients in the voucher condition will attend more psychiatric sessions, which will lead to greater reductions in psychiatric distress.

DETAILED DESCRIPTION:
Male and female opioid-dependent patients at Addiction Treatment Services with any current psychiatric disorder (N = 100) will be randomly assigned to one of two psychiatric service conditions: 1) reinforced on-site integrated care (ROIC), with voucher incentives contingent on attending weekly psychiatric sessions; or 2) standard on-site integrated care (SOIC). Participants in both conditions will receive access to the same schedule and range of psychiatric and substance abuse treatment services. Participants will be assessed for 3-months post-randomization to determine rates of service utilization and adherence to psychiatric care, changes in scope and severity of psychiatric and psychosocial problems, and rates of drug use and treatment retention. Positive findings would have considerable heuristic and health care policy and practice implications. The entire study, including dissemination of the major findings at a national meeting and submission of the first manuscript, is designed to be completed within 2-years.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Voluntarily seeking psychiatric treatment
* Meets DSM-IV criteria for opiate dependence
* Meets FDA/CSAT guidelines for methadone maintenance
* Meets DSM-IV criteria for at least one current psychiatric disorder

Exclusion Criteria:

* Pregnancy
* Onset or acute exacerbation of a medical illness requiring immediate and intense care
* An organic mental disorder (e.g., delirium, dementia)
* Current participation in psychiatric care
* Mandatory psychiatric treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Psychiatric Treatment Adherence | Weekly for 12 weeks
  Patient adherence to all scheduled psychiatric sessions (i.e. individual, group, psychiatrist) will be measured weekly for 12 weeks.
Level of Psychiatric Distress | Every 4-weeks for 12 weeks
  Patients will complete the Addiction Severity Index (ASI) and the SCL-90 every 4-weeks, for 12-weeks, to measure their current levels of psychiatric distress.

SECONDARY OUTCOMES:
Psychiatric Medication Adherence | Every 4-weeks
  Patients will complete a Medication-Taking Scale every 4-weeks to assess their adherence to prescribed psychiatric medications.
Substance Use | Weekly for 12-weeks
  Patients are required to leave weekly urine specimens (for 12-weeks) which are tested for drugs of abuse (opioids, cocaine, benzodiazepines).
Treatment Retention | Weekly for 12-weeks
  The length of time subjects remain in treatment is tracked throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kidorf, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Addiction Treatment Services, Baltimore, Maryland, United States

REFERENCES:
- [Result] Kidorf M, Brooner RK, Gandotra N, Antoine D, King VL, Peirce J, Ghazarian S. Reinforcing integrated psychiatric service attendance in an opioid-agonist program: a randomized and controlled trial. Drug Alcohol Depend. 2013 Nov 1;133(1):30-6. doi: 10.1016/j.drugalcdep.2013.06.005. Epub 2013 Jul 15. PMID 23866988